CLINICAL TRIAL: NCT01177423
Title: Efficiency Evaluation of Intradiploic Intra-osseus Anesthesia Versus Inferior Alveolar Nerve Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2009-08; 2009-A00684-53
Record Dates: First submitted 2009-10-15; First posted 2010-08-09 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Dental Pain
Keywords: restorative odontology; Patients cared in restorative odontology department
MeSH Terms: conditions — Toothache | interventions — Anesthesia, Dental

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Quicksleeper intraosseous anesthesia (Active Comparator): Pulpal and periapical molar and premolar sedation is managed by Quicksleeper intraosseous anesthesia.
  Interventions: Procedure: Dental anesthesia
- Inferior alveolar nerve block (Active Comparator): Pulpal and periapical molar and premolar sedation is managed by inferior alveolar nerve block.
  Interventions: Procedure: Dental anesthesia

INTERVENTIONS:
Procedure: Dental anesthesia — Pulpal and periapical molar and premolar sedation is randomly managed among studied population and Pulp-tester measures anesthesia minute by minute.

SUMMARY:
Management of dental pain emergencies is a challenge for the clinician, particularly when pain is due to endodontic infection.

Tested hypothesis is intradiploic anesthesia is more effective and quicker than inferior alveolar nerve block for mandibular molars anesthesia.

The aim of the study is the evaluation of Quicksleeper efficiency used in first intention versus inferior alveolar nerve block used in most current dental treatment.

DETAILED DESCRIPTION:
Management of dental pain emergencies is a challenge for the clinician, particularly when pain is due to endodontic infection. Failure rate of local anesthesia highly increases with irreversible pulpitis or inflamed periradicular tissue.

Tested hypothesis is intradiploic anesthesia is more effective and quicker than inferior alveolar nerve block for mandibular molars anesthesia (from teeth 35 up to 38 and from 45 up to 48).

The primary aim of the study is the evaluation of Quicksleeper efficiency used in first intention versus inferior alveolar nerve block used in most current dental treatment.

Four clinical situations are evaluated : pulpitis; periapical abcess; pulpal hyperemia; asymptomatic decayed tooth.

Evaluated parameters are : speed of sedation, ability of cure, additional anesthesia needed, total of needles and cartridges used, side effects. Time and validation of complete anesthesia is controlled by pulp tester.

Studied population is patients cared in restorative, endodontics department.

Pulpal and periapical molar and premolar sedation is randomly managed by inferior alveolar nerve block or Quicksleeper intraosseous anesthesia, among studied population (divided in 2 groups of 50 patients). Pulp-tester measures anesthesia minute by minute.

The comparison of study results to bibliography, guidelines and advantages for using mechanical Quicksleeper anesthesia system will be discussed.

ELIGIBILITY:
Inclusion Criteria:

* Irreversible pulpitis on second mandibular premolar or mandibular molars
* Necessity of pulpotomy or pulpectomy

Exclusion Criteria:

* Pregnancy, chest feeding
* Non dental emergency state
* hypersensibility to local anesthesia
* Pheochromocytoma
* Irregularity of cardiac rhythm
* Myocardial infarct in the 6 previous months
* Hepatic porphyria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2009-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the Quicksleeper efficiency used in first intention versus inferior alveolar nerve block used in most current dental treatment. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Herve TASSERY, Principal Investigator — Assistance Publique-Hôpitaux de Marseille
Locations (1):
- Assistance Publique - Hôpitaux de Marseille, Marseille, France